CLINICAL TRIAL: NCT02709083
Title: First-Line Dasatinib or Nilotinib Followed by Response Guided Switch to Imatinib in Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia
Brief Title: Dasatinib or Nilotinib Followed by Imatinib in Patients With Newly Diagnosed, Chronic Phase Chronic Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original principal investigator left institution
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Blum, Acting Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087045; NCI-2016-00162 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3143-16 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myelogenous Leukemia; Chronic Myeloid Leukemia; Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Dasatinib; Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment-dasatinib, nilotinib, imatinib (Experimental): Patients receive dasatinib orally (PO) once a day (QD) or nilotinib PO twice a day (BID) at the discretion of the treating hematologist. Patients achieving either a 1 log reduction at 3 months or a 2 log reduction at 6 months in their breakpoint cluster region-abelson murine leukemia viral oncogene homolog 1 (BCR-ABL1) transcript levels may switch to imatinib mesylate PO QD.
  Interventions: Drug: Dasatinib; Drug: Imatinib Mesylate; Drug: Nilotinib

INTERVENTIONS:
Drug: Dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
Drug: Imatinib Mesylate — Given orally
  Other Names: CGP57148B; Gleevec; Glivec; STI-571
Drug: Nilotinib — Given orally
  Other Names: AMN 107; Tasigna

SUMMARY:
This phase II trial studies how well dasatinib, nilotinib, and imatinib mesylate works in treating patients with newly diagnosed, previously untreated chronic myeloid leukemia in which fewer than 10% of the cells in the blood and bone marrow are blast cells (immature blood cells) (chronic phase). Dasatinib, nilotinib, and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess incidence of major molecular response (MMR) at 12 months.

SECONDARY OBJECTIVES:

I. To assess progression free survival (PFS) at 12 and 24 months.

II. To assess accelerated phase (AP) or blast phase (BP) transformation-free survival at 12 and 24 months.

III. To assess incidence of deep MRs (≥ MR⁴) at 12 months and 24 months.

IV. To assess safety.

V. To assess patient reported outcomes (PRO).

TERTIARY OBJECTIVES:

I. To assess prognostic significance of detecting aberrant myeloid or lymphoid markers on diagnostic bone marrow.

II. To assess ability to enroll subjects who maintain deep molecular remissions in tyrosine kinase inhibitors (TKIs) discontinuation trials.

OUTLINE:

Patients receive dasatinib orally (PO) once a day (QD) or nilotinib PO twice a day (BID) at the discretion of the treating hematologist. Patients achieving either a 1 log reduction at 3 months or a 2 log reduction at 6 months in their breakpoint cluster region-abelson murine leukemia viral oncogene homolog 1 (BCR-ABL1) transcript levels may switch to imatinib mesylate PO QD.

After completion of study treatment, patients are followed up at 2 weeks and then up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated chronic phase chronic myeloid leukemia (CP-CML) (by World Health Organization [WHO] definition) (hydroxyurea permitted up to 7 days prior to enrollment)
* Clinically significant gastrointestinal disease, digestive dysfunction, or surgery that would compromise absorption of oral administration of medications
* Able to give written informed consent and comply with all study visits and procedures

Exclusion Criteria:

* Chronic myeloid leukemia (CML) in AP or BP
* Unable to receive TKI for insurance reasons (uninsurable)
* Refuse or unable to perform telephone or video conferences with research coordinator
* Subjects who are pregnant, breast feeding or sexually active and unwilling to use effective birth control while on treatment with TKI
* Any medical or psychological condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial, poses any additional risk for the subject, or confounds the assessment of the subject

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Started | 7
Completed | 0
Not Completed | 7
Not completed — Original PI left institution | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  Age 20-29 | 2
  Age 30-39 | 3
  Age 40-49 | 0
  Age 50-59 | 0
  Age 60-69 | 1
  Age 70-79 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieve Major Molecular Response (MMR)
Description: Response will be measured by a decrease in fusion transcript or protein resulting from the 9;22 chromosomal translocation responsible for formation of the Philadelphia Chromosome (BCR-ABL1) levels on a logarithmic scale. A 1 log reduction is a drop to below 10%, while a major molecular response (MMR) is defined as a 3 log reduction (0.1%).
Time Frame: At 12 months
Population: Data not collected since trial closed early; original study principal investigator Vamsi Kota, MD, left Emory University.
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Accelerated Phase (AP) or Blast Phase (BP) Free Survival
Description: Survival will be defined as the time from CML diagnosis to the time of transformation to accelerated phase (AP) or blast phase (BP).
Time Frame: The time of CML diagnosis to the time of transformation to AP or BP, assessed up to 24 months
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Patient Reported Outcomes (PRO) Score Extracted From the MD Anderson Symptom Inventory-Chronic Myelogenous Leukemia (CML)
Description: The patient reported outcomes (PRO) score extracted from the MD Anderson Symptom Inventory (MDASI)-Chronic Myelogenous Leukemia (CML) will be determined and intra and inter subject changes will be compared.
Time Frame: Baseline to up to 12 months
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Adverse Events (AEs) Using the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Criteria
Description: Listings of laboratory test results will also be generated, and descriptive statistics summarizing the changes in laboratory tests over time will be presented. Exposure to drug over time will also be summarized. The AE incidence rates, as well as the frequency of occurrence of overall toxicity, categorized by toxicity grades (severity) will be described as obtained from subject forms and subject communications.
Time Frame: Up to 30 days after the end-of-treatment
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of Adverse Events (AEs) Using the Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE v4.03) Criteria
Description: as for outcome 4
Time Frame: Up to 30 days after the end-of-treatment
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) will be defined as the time from CML diagnosis to the time of loss of major molecular response (MMR) or loss of hematologic response.
Time Frame: The time of CML diagnosis to the time of loss of MMR or loss of hematologic response, assessed up to 24 months
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Severity of Adverse Events (AEs) Using the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Criteria
Description: as for outcome 4
Time Frame: Up to 30 days after the end-of-treatment
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

8. Secondary Outcome: The Number of Subjects With Breakpoint Cluster Region-abelson Murine Leukemia Viral Oncogene Homolog 1 (BCR-ABL1) Transcript Levels ≤ Deep Molecular Responses (MR⁴)
Description: Descriptive statistics will summarize the changes in breakpoint cluster region-abelson murine leukemia viral oncogene homolog 1 (BCR-ABL1) testing over time will be presented.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded, concluding 30 days following the last dose of the assigned study treatment.
Arm/Group | Treatment-dasatinib, Nilotinib, Imatinib
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Trial was terminated early due to original study principal investigator Vamsi Kota, MD, leaving Emory University.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02709083/Prot_SAP_000.pdf